CLINICAL TRIAL: NCT00604513
Title: A Theater-Based Obesity Prevention Program for Children
Brief Title: Ready. Set. ACTION! A Theater-Based Obesity Prevention Program for Children
Acronym: RSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0504S69518; R21DK072972 (NIH)
Record Dates: First submitted 2007-12-05; First posted 2008-01-30 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Other: Ready. Set. ACTION! Protocol
- 2 (Sham Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Ready. Set. ACTION! Protocol — The intervention included three components: theater sessions; booster sessions; and family outreach. After-school theater sessions were conducted in the fall in the intervention schools. Sessions included: a "check-in" about changes made over the past week; healthy snacks; a movement component that involved fun and easy activities; and creating/education. Children at intervention schools participated in weekly after-school booster sessions in the winter to further address the behavioral messages addressed during the intervention. Throughout the program, weekly Fun & Fitness packs were sent home to families that included a healthy food with a simple recipe using that food or fitness incentives for the family. There were also two family events: a theater performance, and a reception.
  Arms: 1
Other: Control — The control condition also participated in a theater-based intervention that addressed a health topic unrelated to weight, hand-washing and overall personal hygiene.
  Arms: 2

SUMMARY:
The goal of Ready, Set, ACTION! (RSA) is to test the feasibility of implementing a theater-based after-school program to promote healthy eating, physical activity, and positive body image with children in grades four through six.

DETAILED DESCRIPTION:
The goal of Ready, Set, ACTION! (RSA) is to test the feasibility of implementing a theater-based after-school program to promote healthy eating, physical activity, and positive body image with children in grades four through six. This study, funded by the National Institutes of Health (NIDDK), is a collaboration between the University of Minnesota, Division of Epidemiology and Community Health, Saint Paul Public Schools, and Illusion Theater of Minneapolis. Four participating Saint Paul schools were randomly assigned to receive either a control or intervention after school program led by artists/educators from Illusion Theater. Students in the intervention schools received a fourteen-session curriculum with eight booster sessions, in which they received the following messages: increase fruit, vegetable, and water consumption, decrease soda pop, increase physical activity, and decrease television. Families received nutrition and activity information packets themed for each session. The messages were reinforced by theater education, dance, and music. A play structured around the aforementioned messages that included scene vignettes, choreographed dance, and professionally composed music was developed and rehearsed by the children. In December 2006 the children performed the play for their families at Illusion Theater in downtown Minneapolis. They later performed for their peers at school and again for family and school administrators at the conclusion of the program.

ELIGIBILITY:
Inclusion Criteria:

* 4th-6th grade children at intervention and control schools
* Parent or guardian of participating children

Exclusion Criteria:

* Other ages

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 181 (Actual)
Dates: Start 2006-09; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Program feasibility | One school year

SECONDARY OUTCOMES:
Body Mass Index (BMI) | One school-year
Physical activity | One school-year
Quality of dietary intake | One school-year
Self-efficacy to change eating and physical activity behaviors, improved body image, and improved self-esteem | One school-year
Parental support for healthy eating and physical activity | One school-year

CONTACTS AND LOCATIONS:
Overall Officials: Dianne Neumark-Sztainer, PhD, MPH, RD, Principal Investigator — Division of Epidemiology & Community Health, University of Minnesota